CLINICAL TRIAL: NCT01687179
Title: Targeting Autophagy for the Treatment of TSC and LAM: a Phase I Trial of Hydroxychloroquine and Sirolimus
Brief Title: Safety Study of Sirolimus and Hydroxychloroquine in Women With Lymphangioleiomyomatosis
Acronym: SAIL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Elizabeth Henske, Overall Principal Investigator, Brigham and Women's Hospital
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SAIL-1100; 1ZIAHL002541-21 (NIH)
Record Dates: First submitted 2012-08-02; First posted 2012-09-18 (Estimated); Results first posted 2018-10-11 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: Lymphangioleiomyomatosis
Keywords: LAM; TSC; lymphangioleiomyomatosis
MeSH Terms: conditions — Lymphangioleiomyomatosis | interventions — Sirolimus; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- "Sirolimus" and "Hydroxychloroquine" (Experimental): Subjects will take Sirolimus at an initial dose of 2mg followed by dose adjustment to keep Sirolimus trough levels between 5-15ng/ml consistent with the effective dose in the MILES trial. In addition to Sirolimus subjects will receive Hydroxychloroquine at 200 mg daily for 6 months. Once safety is established at the lower dose ("Sirolimus" and "Hydroxychloroquine" 200 mg), subjects enrolled henceforth will receive Sirolimus and Hydroxychloroquine 400 mg (200 mg twice a day) for 6 months.
  Interventions: Drug: "Sirolimus" and "Hydroxychloroquine" 200 mg; Drug: "Sirolimus" and "Hydroxychloroquine" 400 mg

INTERVENTIONS:
Drug: "Sirolimus" and "Hydroxychloroquine" 200 mg — This will be a phase I dose escalation study of the combination of "Sirolimus" (2 mg adjusted to keep trough levels between 5-15 ng/ml) and "Hydroxychloroquine" 200 mg taken orally daily.
  Other Names: sirolimus(rapamune), hydroxychloroquine (plaquenil)
Drug: "Sirolimus" and "Hydroxychloroquine" 400 mg — Once safety is established with the lower dose, (Sirolimus and Hydroxychloroquine 200 mg), subjects will receive Sirolimus 2 mg (adjusted to keep trough levels between 5 to 15 ng/ml) and hydroxychloroquine 200 mg twice a day.
  Other Names: Sirolimus (Rapamune), Hydroxychloroquine (plaquenil)

SUMMARY:
Specific Aim 1: To investigate whether, in Lymphangioleiomyomatosis (LAM) patients, the combination of sirolimus and hydroxychloroquine is safe and well tolerated

Specific Aim 2: To investigate whether, in LAM patients, 6 months of combination therapy with sirolimus and hydroxychloroquine results in improvement of indicators of disease, and whether the gains are sustained after stopping therapy.

Specific Aim 3: To investigate the potential role of a LAM-specific peripheral blood signature to predict rates of disease progression and determine responsiveness to combination therapy.

This will be a phase I dose escalation study of the combination of sirolimus (2 mg adjusted to keep trough levels between 5-15 ng/ml) and hydroxychloroquine (200 mg or 400 mg) taken orally daily. Up to 18 adult women with LAM will be enrolled.

DETAILED DESCRIPTION:
This will be a phase I dose escalation study of the combination of sirolimus (2 mg adjusted to keep trough levels between 5-15 ng/ml) and hydroxychloroquine (200 mg or 400 mg) taken orally daily for 6 months. The study is to be conducted at 2 sites. Up to 18 adult women with LAM will be enrolled, and each recruiting site will recruit between 8-12 subjects. The protocol will use the following eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Female age 18 or older
* Ability to give informed consent
* Diagnosis of LAM as defined as typical cystic change on CT plus:

  * biopsy or cytology of any tissue demonstrating LAM
  * angiomyolipoma, chylothorax, lymphangioleiomyoma, or tuberous sclerosis
  * serum VEGFD greater or equal to 800pg/ml
* Post-bronchodilator FEV1 equal or less than 80% of predicted or DLCO equal equal or less than 70% of predicted, or RV > 120% of predicted at baseline
* Women of childbearing potential must agree to use 2 forms of barrier contraception during and for 8 weeks after the last dose of medication.

Exclusion Criteria:

* History of intolerance of mTOR inhibitors
* History of intolerance to hydroxychloroquine
* History of severe psoriasis
* History of porphyria cutanea tarda
* Uncontrolled intercurrent illness
* Pregnant, breast feeding, or plan to become pregnant in the next year
* Inadequate contraception
* Significant hematological or hepatic abnormalities
* Use of an investigational drug within 30 days of study start
* Inability to attend scheduled clinic visits
* Inability to perform PFTs
* Creatinine > 2.5mg/dL
* Recent pneumothorax within 8 weeks of screening
* History of malignancy in the last 2 years other than basal cell skin cancer
* Use of estrogen containing medication within 30 days of screening
* Abnormal G6PD levels at baseline
* Preexisting maculopathy or retinopathy
* Preexisting myopathy
* Currently taking doxycycline, metformin, lupron, simvastatin
* Unable to undergo CT or MRI
* History of seizure within last year
* Hepatitis B, C, HIV positive serology
* Use of alternative medical therapies for LAM for at least 6 weeks prior to study participation
* History of myocardial infarct, angina, or stroke related to atherosclerosis
* History of cardiomyopathy
* Previous lung transplant
* Surgery (involving entry into a body cavity or requiring 3 or more stitches) within 2 months of initiation of study drug
* Uncontrolled cholesterol > 350mg/dL, triglycerides > 400mg/dL

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth P Henske, MD, Principal Investigator — Brigham and Women's Hospital; Joel Moss, MD, PhD, Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang Y, El-Chemaly S, Taveira-Dasilva A, Goldberg HJ, Bagwe S, Rosas IO, Moss J, Priolo C, Henske EP. Alterations in Polyamine Metabolism in Patients With Lymphangioleiomyomatosis and Tuberous Sclerosis Complex 2-Deficient Cells. Chest. 2019 Dec;156(6):1137-1148. doi: 10.1016/j.chest.2019.05.038. Epub 2019 Jul 9. PMID 31299246
- [Derived] Lamattina AM, Taveira-Dasilva A, Goldberg HJ, Bagwe S, Cui Y, Rosas IO, Moss J, Henske EP, El-Chemaly S. Circulating Biomarkers From the Phase 1 Trial of Sirolimus and Autophagy Inhibition for Patients With Lymphangioleiomyomatosis. Chest. 2018 Nov;154(5):1070-1082. doi: 10.1016/j.chest.2018.08.1029. Epub 2018 Aug 23. PMID 30144422
- [Derived] El-Chemaly S, Taveira-Dasilva A, Goldberg HJ, Peters E, Haughey M, Bienfang D, Jones AM, Julien-Williams P, Cui Y, Villalba JA, Bagwe S, Maurer R, Rosas IO, Moss J, Henske EP. Sirolimus and Autophagy Inhibition in Lymphangioleiomyomatosis: Results of a Phase I Clinical Trial. Chest. 2017 Jun;151(6):1302-1310. doi: 10.1016/j.chest.2017.01.033. Epub 2017 Feb 10. PMID 28192114

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirolimus and Hydroxychloroquine 200 mg: This will be a phase I dose escalation study of the combination of sirolimus (2 mg adjusted to keep trough levels between 5-15 ng/ml) and hydroxychloroquine 200 mg taken orally daily.
- Sirolimus and HydroxyChloroquine 400 mg: Once safety is established with the lower dose, (Sirolimus and Hydroxychloroquine 200 mg), subjects will receive Sirolimus 2 mg (adjusted to keep trough levels between 5 to 15 ng/ml) and hydroxychloroquine 200 mg twice a day.
Period: Overall Study
Arm/Group | Sirolimus and Hydroxychloroquine 200 mg | Sirolimus and HydroxyChloroquine 400 mg
Started | 3 | 10
Completed | 2 | 6
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Population: 1 subject failed to qualify for the study at the screening visit. Since the subject had signed consent, we considered the participant to be enrolled on the study.
Groups:
- Sirolimus and Hydroxychloroquine: Subjects will take sirolimus at an initial dose of 2mg followed by dose adjustment to keep sirolimus trough levels between 5-15ng/ml consistent with the effective dose in the MILES trial. In addition to sirolimus subjects will receive hydroxychloroquine at 200 mg daily or twice a day for 6 months, depending on time of enrollment into the study, following a standard phase I dose escalation.
  sirolimus and hydroxychloroquine: This will be a phase I dose escalation study of the combination of sirolimus (2 mg adjusted to keep trough levels between 5-15 ng/ml) and hydroxychloroquine (200 mg or 400 mg) taken orally daily.
Arm/Group | Sirolimus and Hydroxychloroquine
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] — Population: 1 subject screen failed.
  years
    number analyzed (Participants) | 13
    (all) | 49 [40 to 65]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 subject screen failed.
  Participants
    number analyzed (Participants) | 13
    Female | 13
    Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 1 subject screen failed.
  Participants
    number analyzed (Participants) | 13
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 12
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: 1 subject screen failed.
  Participants
    United States: number analyzed (Participants) | 13
    United States | 13
Post-Menopause [Count of Participants; unit: Participants] — Population: 1 subject screen failed.
  Participants
    number analyzed (Participants) | 13
    (all) | 6
Pneumothorax [Count of Participants; unit: Participants] — Population: 1 subject screen failed.
  Participants
    number analyzed (Participants) | 13
    (all) | 9
Angiomyolipoma [Count of Participants; unit: Participants] — Population: 1 subject screen failed.
  Participants
    number analyzed (Participants) | 13
    (all) | 2
Tuberous Sclerois (TSC)- Lymphangioleiomyomatosis (LAM) [Count of Participants; unit: Participants] | 0
Lung Biopsy [Count of Participants; unit: Participants] — Population: 1 subject screen failed.
  Participants
    number analyzed (Participants) | 13
    (all) | 8
Chylothorax [Count of Participants; unit: Participants] — Population: 1 subject screen failed
  Participants
    number analyzed (Participants) | 13
    (all) | 1
6 minute walk distance (6MWD) (m) [Mean (Standard Deviation); unit: m] — Population: 1 subject screen failed.
  m
    number analyzed (Participants) | 13
    (all) | 442 (103)
St. George's Respiratory Questionnaire (SGRQ) [Mean (Standard Deviation); unit: units on a scale] — The Saint George's Respiratory Questionnaire (SGRQ) is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scores range from 0 to 100, with higher scores indicating more limitations. Population: 1 subject screen failed.
  units on a scale
    number analyzed (Participants) | 13
    (all) | 43.8 (19.2)
Log VEGF-D (Veascular Endothelial Growth factor) [Mean (Standard Deviation); unit: log(pg/ml)] — Population: 1 subject screen failed.
  log(pg/ml)
    number analyzed (Participants) | 13
    (all) | 3.11 (0.33)
FEV1 [Mean (Standard Deviation); unit: Litres] — Population: 1 Subject Screen failed.
  Litres
    number analyzed (Participants) | 13
    (all) | 1.6 (0.7)
FEV1 (%) [Mean (Standard Deviation); unit: Percent predicted] | 59 (21)
FVC (L) [Mean (Standard Deviation); unit: Litres] — Population: 1 subject screen failed.
  Litres
    number analyzed (Participants) | 13
    (all) | 2.8 (0.7)
FVC (%) [Mean (Standard Deviation); unit: Percent predicted] — Population: 1 Subject Screen failed.
  Percent predicted
    number analyzed (Participants) | 13
    (all) | 81 (16)
DLCO (ml/min/mmhg) [Mean (Standard Deviation); unit: ml/min/mmhg] — Population: 1 Subject screen failed.
  ml/min/mmhg
    number analyzed (Participants) | 13
    (all) | 9.8 (3.1)
DLCO (%) [Mean (Standard Deviation); unit: percent predicted] — Population: 1 Subject screen failed.
  percent predicted
    number analyzed (Participants) | 13
    (all) | 43 (15)

OUTCOME MEASURES:

1. Primary Outcome: Safety of Combination Therapy With Sirolimus and Hydroxychloroquine in LAM Patients
Description: The Primary endpoint of this study was safety. Safety was assessed based on the adverse events and serious adverse events that occurred in these patients when they were on this combination therapy. Percentage of adverse events in each system at a dose was calculated from the total adverse events at that dose. Subjects were closely monitored and adverse events were classified and graded according to the "Common Terminology Criteria for Adverse Events, (CTCAE) Version 4.0".
Time Frame: 48 weeks
Measure: Number; unit: Percentage of adverse events
Groups:
- Sirolimus and Hydroxychloroquine 200 mg: This will be a phase I dose escalation study of the combination of sirolimus (2 mg adjusted to keep trough levels between 5-15 ng/ml) and hydroxychloroquine 200 mg taken orally daily. Safety of the drug combination was assessed by the occurrence of adverse events in these 3 patients.
- Sirolimus and Hydroxychloroquine 400 mg: Once safety is established with the lower dose, (Sirolimus and Hydroxychloroquine 200 mg), subjects will receive Sirolimus 2 mg (adjusted to keep trough levels between 5 to 15 ng/ml) and hydroxychloroquine 200 mg twice a day. Safety of this dose was assessed by the occurrence of adverse events in these 10 patients.
Arm/Group | Sirolimus and Hydroxychloroquine 200 mg | Sirolimus and Hydroxychloroquine 400 mg
Number analyzed (Participants) | 3 | 10
Percentage of adverse events
  Cardiac Disorders | 2.27 | 1.11
  Eye Disorders | 0 | 1.11
  GI Disorders | 18.18 | 22.22
  General Disorders, Administration site condistions | 18.18 | 6.67
  Immune System disorders | 0 | 0.56
  Infections and infestations | 15.91 | 8.33
  Injury, poisoning, procedural complications | 0 | 0.56
  Investigations | 6.82 | 20
  Metabolism and nutrition disorders | 0 | 3.33
  Musculoskeletal, connective tissue disorders | 0 | 4.44
  Nervous system disorders | 4.55 | 5.00
  Psychiatric disorders | 0 | 0.56
  Renal and urinary disorders | 0 | 7.78
  Reproductive system and breast disorder | 6.82 | 1.11
  Respiratory, thoracic, mediastinal disorders | 2.27 | 9.44
  Skin and Subcutaneous disorders | 25.0 | 6.11
  Vascular disorders | 0 | 1.67

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Sirolimus and Hydroxychloroquine 200 mg | Sirolimus and Hydroxychloroquine 400 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/10
Other Adverse Events (participants affected / at risk) | 3/3 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus and Hydroxychloroquine 200 mg (N=3) | Sirolimus and Hydroxychloroquine 400 mg (N=10)
radiculitis (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirolimus and Hydroxychloroquine 200 mg (N=3) | Sirolimus and Hydroxychloroquine 400 mg (N=10)
Rash/ Acne (Skin and subcutaneous tissue disorders) | 3 | 5
Abnormal Investigations (Investigations) | 1 | 6
Diarrhea (Gastrointestinal disorders) | 2 | 6
Oral Mucositis (Gastrointestinal disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No